CLINICAL TRIAL: NCT06954519
Title: Impact of Mental Imagery of Cognitive Neonatal Resuscitation Aid Compared to Simple Reading on the Non-technical Skills of Anaesthesia Residents Six Months After Initial Training: a Randomized Study
Brief Title: Impact of Mental Imagery on the Non-technical Skills of Anaesthesia Residents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reims University hospital (Other)
Responsible Party: Principal Investigator, Michelet Daphne, Clinical Professor, Reims University hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Mental imagery study
Record Dates: First submitted 2025-03-27; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: no Condition is Studied; the Focus of the Study is the Impact of Mental Imagery on Non Technical Skills of Medical Students
Keywords: mental imagery; cognitive aid; neonatal resuscitation; simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Imagery (Experimental): Participant of the mental imagery group will have a specific training during the initial training and will repeat the mental imagery regularely during the 6 months (timing of repetition guided by messages sended by investigator)
  Interventions: Other: Mental imagery
- Classical reading (Active Comparator): Participant of the control group will have no specific training during the initial training, only presentation of the cognitive aid. They will also repeat the reading of the cognitive aid regularely during the 6 months (timing of repetition guided by messages sended by investigator)
  Interventions: Other: Cognitive aid reading

INTERVENTIONS:
Other: Mental imagery — The principle of guided mental imagery and helping students to mentally represent the key stages of a process, using an animated slideshow full of evocative elements, which we created specifically for this study. The mental imagery will be repeated by the students several times independently until the evaluation simulation at 6 months based on reminders via messages from investigators.
  Arms: Mental Imagery
Other: Cognitive aid reading — Participants of the control group will only read the cognitive aid on neonatal resuscitation at the same intervalls than the experimentation group
  Arms: Classical reading

SUMMARY:
The goal of this randomized trial is to learn if mental imagery works to improve non technical skills in residents. It will also learn about knowledge and technical skills. The main questions it aims to answer are:

Does mental imagery of a cognitive aid improve non technical skills of residents ? Does mental imagery of a cognitive aid improve technical skills and knowledge of residents ?

The invastigators will compare repeated mental imagery to repeated simple reading of a cognitive aid to see if mental imagery works to train non technical skills.

Participants will:

* participate in an initial training on neonatal resuscitation
* be randomized in two groups: mental imagery or simple reading
* Repeat training according to the group with predefined intervalls during 6 months
* be evaluated 6 months after the initial training

DETAILED DESCRIPTION:
Non-technical skills, such as stress management, decision-making, communication and leadership, are crucial in anaesthesia and intensive care, particularly in emergency situations where technical performance alone is not enough. Mental imagery training used in the fields of sport and surgery could play a key role in improving these skills in future doctors.

A recent study showed that mental imagery training led to better non-technical skills among first-year anaesthesia residents in simulation of a cardiopulmonary resuscitation case (article currently being reviewed).

This study compared mentalisation with reminders at predefined intervals in the intervention group with no reminders to read the cognitive aid in the control group. In addition, cardiopulmonary arrest is a well-known subject for students and initial knowledge was not assessed beforehand.

This new clinical trial aims to evaluate the impact of mental imagery on the non-technical skills of anaesthesia and intensive care residents following initial training in neonatal resuscitation with a full-scale simulation evaluation at 6 months, in residents with a reminder of mentalisation or rereading of the cognitive aid depending on the group.

1. Objective of the study 2.1 Main objective: Blind video assessment by an expert examiner of the non-technical skills (situational awareness, communication, decision-making, teamwork) of anaesthesia and intensive care residents on a simulated neonatal resuscitation case with the BARS score out of 36 points (9 for the 4 subcategories of non-technical skills).

   2.2 Secondary objectives: Assessment of basic knowledge using an initial knowledge quiz, to be repeated after 6 months.

   Blind video assessment of technical skills by an expert examiner using the NRPE score.

   Assessment of participants' visuospatial abilities using the MIQ-R questionnaire, initially and after 6 months.
2. Methodology 2.1 Study population Interns in anaesthesia and intensive care (DESAR 1, 2, 3 and 4)

   Number of subjects required:

   Assuming a change in the BARS score from 20 (control) to 25 (mentalisation) in line with our previous study, a standard deviation of 4, a risk alpha 5% beta 80% and 0 lost to follow-up, 22 participants (11 per group) are required.

   Randomisation:
   * Experimental group: mentalisation of the ILCOR cognitive aid for neonatal resuscitation at predefined intervals
   * Control group: simple reading of the ILCOR cognitive aid for neonatal resuscitation at predefined intervals 2.2 Inclusion criteria Anaesthesia and intensive care interns (DESAR 1, 2, 3 and 4) volunteers Signed informed consent 2.3 Exclusion criteria Refusal to participate in the study 2.4 Intervention
   * Both groups will complete an initial knowledge questionnaire and the MIQR questionnaire, then receive initial neonatal resuscitation training based on a theoretical course followed by practical workshops and simulation.
   * The experimental group will receive guided mentalisation based on ILCOR cognitive aids for neonatal resuscitation. Regular reminders of mentalisation will be given over a period of 6 months before the final evaluation. Adherence to mental rehearsals will be verified.
   * The control group will receive ILCOR cognitive aids for neonatal resuscitation. Regular reminders to read the cognitive aid will be given over a period of 6 months before the final evaluation. Adherence to the reminders will be verified.
3. Statistical analysis Mann-Whitney U test for independent samples Statistical analyses performed using SPSS software. Significance level set at p < 0.05
4. Ethical considerations Informed consent obtained from all participants, guaranteeing their right to confidentiality and anonymity.
5. Study schedule 27 March: randomisation and inclusion of participants in two groups. 27 March: knowledge questionnaire and MIQR, theory lesson with presentation of cognitive aid, handling of equipment, MCE, IOT, guided mentalisation for the mentalisation group.

   April-October: reminder messages at predefined intervals for both groups October: final evaluation in individual simulation over a 10-minute period, filmed, scenario to be defined, knowledge questionnaire and MIQR. Evaluation of the videos by 2 experts not involved in the study.
6. Conclusion The objective of this study is to analyse whether regular training using mental imagery can improve the non-technical skills of anaesthesia and intensive care interns compared to reading a cognitive aid, and thus potentially increase the effectiveness of medical teams in emergency situations.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia residents in 1, 2, 3 o 4 year of training and volunteers

Exclusion Criteria:

* Residents not volunteer

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Behaviorally Anchored Rating Scale (BARS) | 6 months
  Evaluation of Non-Technical Skills of anesthesia residents' (Originally published in Watkins et al., Simul in Healthc 2017). From 1 to 36 points. Better score means better skills

SECONDARY OUTCOMES:
Neonatal Resuscitation Performance Evaluation (NRPE) scale | 6 months
  Score evaluationg the different phases of neonatal resuscitation (A, B, C). Score on 20 points. Better score means better management.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Reims, Reims, Grand Est
  - CHU de Reims, Reims

IPD SHARING:
Plan to Share IPD: No